CLINICAL TRIAL: NCT01967797
Title: Implementation and Validation of the "5As Framework of Obesity Management" in Primary Care. "5AsT"
Acronym: 5AsT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Edmonton South Side Primary care network (Unknown); Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RES 0014622
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2016-03

CONDITIONS: Overweight and Obesity
Keywords: Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5As Team Intervention (Experimental): The intervention group will participate in an additional 6 month intensive learning collaborative model designed around the 5As of obesity management, but which addresses areas identified as barriers (i.e. weight bias, clinical environment, clinic processes & team based care, mental health, counseling around emotional eating, caregiver fatigue, designing appropriate patient follow-up, and additional topics identified by the professionals). A clinical Champion identified by our partner SSPCN will be available to provide 1:1 support and coaching of the practitioners & teams as needed. The practitioners will work collaboratively to do their own needs assessment, and will identify additional resources or tools that they need to overcome the barriers to weight management in their setting. The research team will use a Practice Facilitation model to provide additional resource and support to the change process for the practitioners.
  Interventions: Behavioral: 5As Team Intervention
- Control (No Intervention): Though the controls will have knowledge of the '5A's of Obesity Management', they will not be receiving 5As Team Intervention.

INTERVENTIONS:
Behavioral: 5As Team Intervention — The intervention group will participate in an additional 6 month intensive learning collaborative model designed around the 5As of obesity management, but which addresses areas identified as barriers (i.e. weight bias, clinical environment, clinic processes & team based care, mental health, counseling around emotional eating, caregiver fatigue, designing appropriate patient follow-up, and additional topics identified by the professionals). A clinical Champion identified by our partner SSPCN will be available to provide 1:1 support and coaching of the practitioners & teams as needed. The practitioners will work collaboratively to do their own needs assessment, and will identify additional resources or tools that they need to overcome the barriers to weight management in their setting. The research team will use a Practice Facilitation model to provide additional resource and support to the change process for the practitioners.
  Arms: 5As Team Intervention

SUMMARY:
The main goal of this project is to develop, implement and evaluate the 5As Team intervention (5AsT)for healthcare practitioners to improve their weight management patient encounters and improve patient health outcomes. The 5As of Obesity Management suite of tools is a robust, evidence-based approach to weight management, however its implementation and uptake has been heterogeneous in primary care.

This project was co-created by, and will be implemented with, our partners the Southside Primary Care Network (SSPCN). A needs assessment on weight management by the SSPCN revealed the need to change provider practice to increase the number of weight management visits. Despite a robust didactic training session on weight management for all providers, which includes the 5As, the uptake in practice has been highly heterogeneous. Thus, the 5AsT intervention to address the implementation of the 5As of Obesity Management in clinical practice was developed by the collaborative team. The SSPCN consists of 25 autonomous groups of multidisciplinary professionals that provide service to a defined group of patients within the SSPCN.

The 5As Team consists of multidisciplinary providers (Registered Nurse/ Nurse Practitioner, dietician, mental health worker) who work collaboratively. The intervention is a learning collaborative where these 12 different 5AsTs get together to work to address facilitators and barriers to weight management in their settings over a 6 month period. Half of the teams (N=12) will remain as controls and deliver usual care. They serve as a comparison group for the 5AsTs. This mixed methods study's primary outcomes will assess the change in provider practice and the effectiveness of the intervention and implementation.

To assess the impact of 5AsT on patients, we will recruit patients presenting to the central SSPCN programming, We will not intervene directly on patients; we will observe the impact of the 5AsT and SSPCN programming on their health outcomes for a minimum of 6 months, and where possible for 18 months. Data collected includes demographics, weight (BMI), waist circumference, vital signs,and Short Form-12 (SF-12,these measures are routinely measured in the SSPCN), EuroQol-5 dimensions 5 Level (EQ-5D-5L), modified patient assessment of chronic illness (PACIC), and observed adherence to routine clinical care for guideline recommended laboratory monitoring (cholesterol panel, fasting glucose, HbA1c, where appropriate).

DETAILED DESCRIPTION:
Obesity is a public health problem as it is associated with many co-morbidities, decreased life expectancy and high health care costs. In 2008, prevalence of obesity and overweight, combined, in Canada was 62.1%. Supported by Canadian Institute of Health Research (CIHR) and Public Health Agencies of Canada Innovation strategy, the Canadian Obesity Network developed a novel tool for obesity counseling and management in primary care settings know as the "5As of Obesity Management". However, despite current dissemination strategies and extensive provider education in the 5As, the uptake of current practices for weight management has been inconsistent. Evidence suggests that treating obesity can reduce the incidence of a number of chronic diseases, and that obesity is not effectively managed in our current health care system.This project was co-created by, and will be implemented with, our partners the Southside Primary Care Network (SSPCN).

The main goal of this project is to develop and evaluate a pragmatic intervention called the 5As Team Intervention(5AsT) which acts on health professionals, forming them into a 6 month learning collaborative that undergoes an iterative, action based process to address facilitators and barriers to weight management.

Primary Objective:

Increase the number of weight management visits conducted by SSPCN Registered Nurses/Nurse Practitioners (RN/NPs).

Primary questions:

1. Does the 5As Team (5AsT) intervention affect the number of weight management visits conducted by SSPCN practitioners (RN/NP) in their SSPCN practice?
2. Under what circumstances does the 5AsT intervention affect the number of weight management visits conducted by the SSPCN practitioners?
3. Are changes in weight management visit rates sustained following the intervention period?
4. What is the impact of implementation of 5AsT on practice level outcomes - on unique 5As Teams and the SSPCN?

Secondary Objective:

To evaluate the impact of SSPCN weight management programming, with and without this 5AsT intervention, on patient important outcomes including: weight (BMI), blood pressure, self reported health status (EQ5D,SF-12), and patient-reported measures of chronic disease management for obesity (modified PACIC), as well as completion of appropriate laboratory studies (HbA1c for diabetics, fasting glucose, and cholesterol panel for age>40).

Design: This is a mixed methods, pragmatic cluster randomized trial in regular practice. The quantitative portion focuses on provider weight management visits, and patient-important outcomes above. For the patient study, 2 primary patient outcomes the study is powered for are BMI and SF-12, the remainder above are secondary patient outcomes. The qualitative portion seeks to understand the implementation process and the efficacy of the 5AsT intervention. Practitioners affiliated with different clinical groups will be randomized to intervention or control. All practitioners receive a robust didactic training program in weight management. The intervention group practitioners will participate in a 6 month 5AsT learning collaborative to address barriers to implementation of effective weight management strategies based upon the 5As of Obesity Management tool kit. Interested patients presenting to the central SSPCN programming will be recruited to participate in the study. There is no study intervention on the patients; the study will only observe how they are doing on their weight management journey in the SSPCN - whether they come from an intervention or control practice group. We will conduct a rigorous qualitative analysis of the intervention process using numerous qualitative tools to assess both the intervention itself and participant views. A qualitative plan has been created that outlines the use of field notes, focus groups and interviews to collect data and the use of Thematic Analysis and Nvivo software for analysis.

Intervention: The 5As Team (5AsT) Program intervention in this study is based on behavior change theory. The Teams are groups of SSPCN practitioners (RN/NP, Social work, Registered Dietitian) who practice collaboratively in the community (N=25). The intervention group (N=12 teams) will participate in an additional 6 month intensive learning collaborative model designed around the 5As of obesity management, but which addresses areas identified as barriers (i.e. weight bias, clinical environment, clinic processes & team based care, mental health, counseling around emotional eating, caregiver fatigue, designing appropriate patient follow-up, and additional topics identified by the professionals). A clinical Champion identified by our partner SSPCN will be available to provide 1:1 support and coaching of the practitioners & teams as needed. The practitioners will work collaboratively to do their own needs assessment, and will identify additional resources or tools that they need to overcome the barriers to weight management in their setting. The research team will use a Practice Facilitation model to provide additional resource and support to the change process for the practitioners.

Setting: The SSPCN is one of the largest Primary Care Networks (PCN) in Alberta, which serves an ethnically and socially diverse population from 45 community family practices. The SSPCN centralizes programs that are not available at independent family practices. Also, each primary care center has a SSPCN team of personnel who reports directly to the SSPCN, and are responsible for delivering services to patients from that patient catchment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years
* BMI ≥ 25
* Enrolling in PCN programs for overweight/ obesity or depression able and willing to give written informed consent in English

Exclusion Criteria:

* Children and pregnant women
* Patients whose obesity is co-managed by an obesity specialist or tertiary care center
* Patients who are unable to participate in regular clinic visits or programs due to geographic, social or physical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Number of weight management visits/ practitioner Full Time Equivalent(FTE) | Data will be collected monthly and analyzed at 6, 12 and 18 Months
  PROVIDER INTERVENTION STUDY- This is routine operational data collected by the SSPCN on all encounters conducted by all practitioners. Providers are blinded to the outcome measure.
Change in BMI | 3,6,12,and 18 month where possible
  PATIENT STUDY - Primary outcome measure. All patients receive SSPCN health courses. This measure compares patients from the 5AsT clinics and the control clinics to see whether they have greater weight loss, and more success in sustained weight management. This will also be assessed by the number of interactions they have for weight management over the time frame.
Change in Self-reported health measures-SF12 | 3,6,12 months and 18 months where possible
  PATIENT STUDY-All patients receive central SSPCN health programming. This compares those from 5AsT Team clinics with those from control clinics to see whether they have greater self-reported health measures and more success with sustained improvement. This will also be assessed by the number of interactions they have for weight management over the time frame.

SECONDARY OUTCOMES:
Change in Self-reported health measures- EQ5D | 3,6,12 months and 18 months where possible
  PATIENT STUDY - In order to account for short term health concerns, we are co-administering the EQ-5D-5L.
Change in PACIC Score | 3 months, 6 months, 12 months, and 18 months where possible
  Patient report of health care providers' management of weight as a chronic medical condition. (modified PACIC score)

OTHER OUTCOMES:
Qualitative Description of the Implementation Process | 12 months
  SSPCN Personnel randomized to the study intervention group will be trained for a 6 month period. During training, there will be collection of field notes, 1:1 interviews and focus groups for consenting practitioners. The data will be analyzed on a weekly basis to identify themes concerning the efficacy of the intervention process and practitioner behavior change. This will be used to continually refine the intervention, and describe how and why it is/not working.
  Following the 12 months (6 month intervention, 6 months of monitoring to assess sustainability) both qualitative and quantitative results will be combined to explore correlation. This will allow for more in-depth exploration of any variation in results.

CONTACTS AND LOCATIONS:
Overall Officials: Arya M Sharma, MD,PhD, Principal Investigator — University of Alberta
Locations (1):
- University Of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Campbell-Scherer DL, Asselin J, Osunlana AM, Ogunleye AA, Fielding S, Anderson R, Cave A, Johnson JA, Sharma AM. Changing provider behaviour to increase nurse visits for obesity in family practice: the 5As Team randomized controlled trial. CMAJ Open. 2019 May 30;7(2):E371-E378. doi: 10.9778/cmajo.20180165. Print 2019 Apr-Jun. PMID 31147378
- [Derived] Luig T, Asselin J, Sharma AM, Campbell-Scherer DL. Understanding Implementation of Complex Interventions in Primary Care Teams. J Am Board Fam Med. 2018 May-Jun;31(3):431-444. doi: 10.3122/jabfm.2018.03.170273. PMID 29743226
- [Derived] Asselin J, Salami E, Osunlana AM, Ogunleye AA, Cave A, Johnson JA, Sharma AM, Campbell-Scherer DL. Impact of the 5As Team study on clinical practice in primary care obesity management: a qualitative study. CMAJ Open. 2017 Apr 26;5(2):E322-E329. doi: 10.9778/cmajo.20160090. PMID 28450428
- [Derived] Ogunleye A, Osunlana A, Asselin J, Cave A, Sharma AM, Campbell-Scherer DL. The 5As team intervention: bridging the knowledge gap in obesity management among primary care practitioners. BMC Res Notes. 2015 Dec 22;8:810. doi: 10.1186/s13104-015-1685-8. PMID 26695407
- [Derived] Campbell-Scherer DL, Asselin J, Osunlana AM, Fielding S, Anderson R, Rueda-Clausen CF, Johnson JA, Ogunleye AA, Cave A, Manca D, Sharma AM. Implementation and evaluation of the 5As framework of obesity management in primary care: design of the 5As Team (5AsT) randomized control trial. Implement Sci. 2014 Jun 19;9:78. doi: 10.1186/1748-5908-9-78. PMID 24947045